CLINICAL TRIAL: NCT02417493
Title: Epinephrine Self-injection and Self-management of Food Allergies
Brief Title: Self-injection and Self-management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Fordham University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 15-0140; 02662242 - 4606 (Other Grant/Funding Number: EMPOWER Program, Mount Sinai Hospital)
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-06

CONDITIONS: Food Allergy
Keywords: Food allergy; self-management; epinephrine self-injection; ntervention; adolescents
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simulation of Epinephrine Self-Injection (Experimental): The patient will self-inject an empty syringe into his/her thigh simulating a self-injection of epinephrine during a routine outpatient visit to the allergist.
  Interventions: Behavioral: Simulation of epinephrine self-injection
- Control Group (No Intervention): The patient will be encouraged to speak to their physician about self-injection, but will not undergo the self-injection protocol during a routine outpatient visit to the allergist.

INTERVENTIONS:
Behavioral: Simulation of epinephrine self-injection
  Arms: Simulation of Epinephrine Self-Injection

SUMMARY:
The purpose of the present study is to determine if asking adolescent patients (ages 13-17) to self-inject an empty syringe into their thigh during routine clinic visits results in increased reported comfort with self-injection, reduced anxiety regarding self-injection and food allergy management for both patient and caregiver(s), and in greater perceived likelihood of epinephrine self-injection, in the event of an emergency.

DETAILED DESCRIPTION:
The purpose of the present study is to determine if asking adolescent patients (ages 13-17) to self-inject an empty syringe into their thigh during routine clinic visits results in increased reported comfort with self-injection, reduced anxiety regarding self-injection and food allergy management for both patient and caregiver(s), and in greater perceived likelihood of epinephrine self-injection, in the event of an emergency. Forty participants, in total, will be recruited during routine visits to an outpatient allergy clinic. Half of all participants will be randomized to the behavioral self-management intervention; whereby patients will insert a needle attached to an empty syringe into their thigh (simulating an injection of epinephrine); the other half of participants will be randomized to the control condition, and will be encouraged to speak to their physician about self-injection, but will not undergo the self-injection protocol. Prior to randomization, baseline measures will be collected on patient's comfort with epinephrine self-injection. Following the self-injection protocol and/or the discussion of self-injection with the physician, all participants will complete immediate post-intervention questionnaires at clinic about comfort with self-injection, health care management and anxiety. One month following the clinic visit, all patients will be sent a follow-up questionnaire that will include items identical to the ones completed at immediate post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen in the outpatient clinic and their caretakers (no inpatients).
* Patients must have been diagnosed with food allergy and previously prescribed self-injectable epinephrine.
* Patients between the ages of 13-17 years old.
* Parent consent and child assent.

Exclusion Criteria:

* Patients and caregiver(s) who have been diagnosed with cognitive barriers that prevent them from understanding the study, as determined by either: a previously diagnosed mental retardation or inability to repeat the study protocol at the time of consent.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Child comfort with epinephrine self-injection | Day 1
  Immediate pre-post differences within the intervention group in the score obtained on a child-reported "comfort with self-injection" questionnaire.

SECONDARY OUTCOMES:
Child likelihood of epinephrine self-injection | Day 1
  Immediate pre-post differences within the intervention group in the score obtained on a child-reported likelihood of self-injection questionnaire.
Parent report of child comfort with epinephrine self-injection | Day 1
  Immediate pre-post differences within the intervention group in the score obtained on a parent-reported "child's comfort with self-injection" questionnaire.
Child comfort with epinephrine self-injection | 1 month post-intervention
  Immediate post-1 month post differences between groups in the score obtained on a child-reported "comfort with self-injection" questionnaire.
Parent report of child comfort with epinephrine self-injection | 1 month post-intervention
  Immediate post- 1 month post differences between groups in the score obtained on a parent-reported "child's comfort with self-injection" questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Shemesh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Jaffe Food Allergy Institute, New York, New York, United States